CLINICAL TRIAL: NCT06132542
Title: Autologous Adipose Derived Mesenchymal Stromal Cell Transplantation in Patients With Idiopathic or Drug Induced Premature Ovarian Failure
Brief Title: Autologous ADMSC Transplantation in Patients With POI
Acronym: ADMSC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongolian National University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Batsuren Choijamts, Teacher, Mongolian National University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23/035
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Open label study
  Interventions: Biological: stem cell therapy

INTERVENTIONS:
Biological: stem cell therapy — The fat derived stem cell will be transplanted by a reproductive gynecologist who does routine ovarian puncture.
  Other Names: fat derived stem cell

SUMMARY:
The primary ovarian insufficiency (premature ovarian failure, premature ovarian insufficiency, premature menopause) is a hypergonadotropic hypogonadism, that failure of the ovarian function in woman younger than 40 years. Fat derived stem cells are mainly mesenchymal stem cells and found to be effective treatment in joint and bone regeneration.

We are planning to investigate the effectiveness of adipose stem cell on ovarian tissue regeneration for patients with premature ovarian failure.

DETAILED DESCRIPTION:
The primary ovarian insufficiency (premature ovarian failure, premature ovarian insufficiency, premature menopause) is a hypergonadotropic hypogonadism, that failure of the ovarian function in woman younger than 40 years. Ovary is a important organ of reproduction as well as endocrine organ that secretes estrogen and progesterone to stimulate the endometrium and other organs. The main features of are sex hormone deficiency, amenorrhea, infertility, and elevated serum gonadotropins.

This condition occurs in approximately 1% of women and it has significant psychological and physical consequences in those patients.

The current management involves hormone replacement therapy and infertility treatment using egg donors.

Stem cells are the foundation cells for every organ, tissue, and cell in the body. They are undifferentiated cells that do not yet have specific function. Under proper conditions, they begin to develop into specialized tissue and organs. Fat derived stem cells are mainly mesenchymal stem cells and found to be effective treatment in joint and bone regeneration.

This study is an open-label investigation of the efficacy of injection of autologous adipose derived stem cells into the ovarian stroma of patients with premature ovarian failure. Totally 10 women with POI will be recruited in this study after the written informed consent. Diagnosis will be based mainly on history taking, physical examination, and laboratory investigations. Laboratory investigations will include serum follicle stimulating hormone (FSH), serum estrogen measurement and serum AMH. The typical FSH in POI patients is over 40mIU/ml (post-menopausal range). Subjects will be enrolled based on specific inclusion/exclusion criteria and will be evaluated at regular post-transplant intervals.

The fat derived stem cell will be transplanted by a reproductive gynecologist who does routine ovarian puncture. Subjects will be monitored frequently for a total of one year after ADSCs injection. For the safety of patients, the stem cell will be injected in one ovary only and the other ovary will be spared.

Sample of 150-250 ml aspirated from the fat will be processed according to the manufacturers guide and totally 5 million of ADSCs will be injected into the ovaries under guidance of transvaginal sonography. Endometrial fractional biopsy will be taken, stained with H&E stain. Participants will be followed up monthly for a period of 6 months by hormonal (FSH, LH, E2, AMH), clinical (resuming menstruation), US (folliculometry).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Female over the age of 18
* Diagnosis of premature ovarian insufficiency: At least two menopausal FSH levels (≥ 40 IU/L) and/or Primary or secondary amenorrhea at least for 3-6 months OR Diagnosis of low ovarian reserve defined as: AMH < _0.42 ng/ML & FSH >20 IU/L, and/or failure of prior attempts of assisted reproductive techniques due to limited ovarian response (poor responder).
* Presence of at least one ovary
* Acceptable uterine anatomy (by any clinically and/or imaging acceptable methods)
* Normal thyroid function as evidence by normal serum Thyroid Stimulating Hormone (TSH) levels.
* Agree to report any pregnancy to the research staff immediately.
* Willing and able to comply with study requirements and follow up instructions.

Exclusion Criteria:

* Has a history of, or evidence of current gynecologic malignancy within the past three years
* Presence of adnexal masses indicating the need for further evaluation
* Major mental health disorder that precludes participation in the study
* Active substance abuse or dependence
* Current or recent (within the past 2 weeks) use of the following medications: Oral or systemic corticosteroids, Hormones (estrogen, progestins, oral contraceptives), Danazol, anticoagulants, herbal or botanical supplements with possible hormonal effects. Washout will be allowed.
* Type I or Type II diabetes mellitus, or if receiving antidiabetic medications
* Known significant anemia (Hemoglobin <8 g/dL).
* Untreated deep venous thrombosis, and/or pulmonary embolus
* Untreated cerebrovascular disease
* Known heart disease (New York Heart Association Class II or higher).
* Known Liver disease (defined as Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT)>2 times normal, or total bilirubin >2.5 mg/dL).
* Known Renal disease (defined as Blood urea nitrogen (BUN)>30 mg/dL or serum creatinine > 1.6 mg/dL).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Resumption of menses (12 months) | 12 months
  regular 25-45 day cycle menses, with 2-5 day bleeding.
Improved clinical hormone levels. | 12 months
  FSH 4.7 to 21.5 mIU/mL (4.5 to 21.5 IU/L)

SECONDARY OUTCOMES:
Achievement of pregnancy | 12 months
  A transvaginal ultrasound confirmation of gestational sac The hCG levels have reached between 1,000 - 2,000 mIU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Batsuren Choijamts, Ph.D, Principal Investigator — Mnums
Locations (1):
- Mongolian National University of Medical Science, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Golezar S, Ramezani Tehrani F, Khazaei S, Ebadi A, Keshavarz Z. The global prevalence of primary ovarian insufficiency and early menopause: a meta-analysis. Climacteric. 2019 Aug;22(4):403-411. doi: 10.1080/13697137.2019.1574738. Epub 2019 Mar 4. PMID 30829083
- [Result] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- [Result] Howard-Anderson J, Ganz PA, Bower JE, Stanton AL. Quality of life, fertility concerns, and behavioral health outcomes in younger breast cancer survivors: a systematic review. J Natl Cancer Inst. 2012 Mar 7;104(5):386-405. doi: 10.1093/jnci/djr541. Epub 2012 Jan 23. PMID 22271773
- [Result] Baber RJ, Panay N, Fenton A; IMS Writing Group. 2016 IMS Recommendations on women's midlife health and menopause hormone therapy. Climacteric. 2016 Apr;19(2):109-50. doi: 10.3109/13697137.2015.1129166. Epub 2016 Feb 12. PMID 26872610
- [Result] Anderson RA, Mansi J, Coleman RE, Adamson DJA, Leonard RCF. The utility of anti-Mullerian hormone in the diagnosis and prediction of loss of ovarian function following chemotherapy for early breast cancer. Eur J Cancer. 2017 Dec;87:58-64. doi: 10.1016/j.ejca.2017.10.001. Epub 2017 Nov 5. PMID 29117576
- [Result] Bidet M, Bachelot A, Bissauge E, Golmard JL, Gricourt S, Dulon J, Coussieu C, Badachi Y, Touraine P. Resumption of ovarian function and pregnancies in 358 patients with premature ovarian failure. J Clin Endocrinol Metab. 2011 Dec;96(12):3864-72. doi: 10.1210/jc.2011-1038. Epub 2011 Oct 12. PMID 21994953
- [Result] Sauer MV. Spontaneous pregnancy in women awaiting oocyte donation. J Reprod Med. 1995 Sep;40(9):630-2. PMID 8576878
- [Result] van Kasteren YM, Schoemaker J. Premature ovarian failure: a systematic review on therapeutic interventions to restore ovarian function and achieve pregnancy. Hum Reprod Update. 1999 Sep-Oct;5(5):483-92. doi: 10.1093/humupd/5.5.483. PMID 10582785
- [Result] Alatab S, Shekarchian S, Najafi I, Moghadasali R, Ahmadbeigi N, Pourmand MR, Bolurieh T, Jaroughi N, Pourmand G, Aghdami N. Systemic Infusion of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells in Peritoneal Dialysis Patients: Feasibility and Safety. Cell J. 2019 Jan;20(4):483-495. doi: 10.22074/cellj.2019.5591. Epub 2018 Dec 12. PMID 30123994
- [Result] Mashayekhi M, Mirzadeh E, Chekini Z, Ahmadi F, Eftekhari-Yazdi P, Vesali S, Madani T, Aghdami N. Evaluation of safety, feasibility and efficacy of intra-ovarian transplantation of autologous adipose derived mesenchymal stromal cells in idiopathic premature ovarian failure patients: non-randomized clinical trial, phase I, first in human. J Ovarian Res. 2021 Jan 6;14(1):5. doi: 10.1186/s13048-020-00743-3. PMID 33407794